CLINICAL TRIAL: NCT06910163
Title: Direct-to-angio Approach From loCal hOspitals Based on a PoInt-of-care bLOod Test for LVO (COPILOT): an Effectiveness Cluster Randomized Crossover Trial
Brief Title: Direct-to-angio Approach From loCal hOspitals Based on a PoInt-of-care bLOod Test for LVO
Acronym: COPILOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juan Vicenty (Other)
Collaborators: University of Puerto Rico (Other); Mennonite Health System (Unknown)
Responsible Party: Sponsor-Investigator, Juan Vicenty, MD, University of Puerto Rico
Organization: University of Puerto Rico (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2410303013
Record Dates: First submitted 2025-03-27; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Acute Stroke
Keywords: Acute Stroke; Ischemic Stroke; LVOne Test; Diagnosis; Large Vessel Occlusion (LVO); Glial Fibrillary Acidic Protein (GFAP); D-dimer
MeSH Terms: conditions — Stroke; Ischemic Stroke; Disease

STUDY DESIGN:
Intervention Model Description: The COPILOT trial, a cluster randomized crossover study within the Sistema de Salud Menonita (SSM) hospital network, evaluates whether early detection of large vessel occlusion (LVO) stroke via a novel blood test accelerates triage-to-thrombectomy time.
  Phase 0 (3 months): Baseline data collection to establish pre-intervention comparisons. Patients receive standard care, and an interim analysis assesses recruitment and study power.
  Phase 1 (12 months): Clusters are randomized to intervention (LVOne test) or control (standard care). Analysts remain blinded, and interim analysis reassesses recruitment and primary outcomes.
  Phase 2 (12 months): Clusters switch roles, enabling within-cluster comparisons. Due to the intervention's nature, participants and staff cannot be blinded.
Who Masked: Outcomes Assessor
Masking Description: The neuro-radiologist(s) who will read patient brain imaging and the expert stroke clinician(s) who will assign a clinical outcome (reference standard) will be blinded to the LVOne test results. Due to the nature of the LVOne and the management implications of a positive test, hospital clinicians will not be blinded to these results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Participants will receive the current diagnostic standard of care.
  Interventions: Diagnostic Test: Diagnostic standard of care
- LVOne Test (Experimental): Participants will receive the LVOne test alongside the current standard of care.
  Interventions: Diagnostic Test: Diagnostic standard of care; Diagnostic Test: LVOne Test

INTERVENTIONS:
Diagnostic Test: Diagnostic standard of care — Participants will receive the diagnostic standard of care: standard laboratory workup, non-contrast brain CT, brain CTA, brain CTP, or brain MRI.
Diagnostic Test: LVOne Test — Participants will receive the LVOne test, which will measure D-dimer and Glial Fibrillary Acidic Protein (GFAP) levels to diagnose acute stroke.
  Arms: LVOne Test

SUMMARY:
Direct-to-angio approach from loCal hOspitals based on a PoInt-of-care bLOod Test for LVO (COPILOT) is a multi-center, prospective, cluster-randomized crossover trial that will evaluate if the triage assessment to thrombectomy puncture time is shorter after performing the LVOne testing compared to current management standards in patients with suspected large vessel occlusion.

DETAILED DESCRIPTION:
The COPILOT trial utilizes a cluster randomized crossover design within the Sistema de Salud Menonita (SSM) hospital network to evaluate if early detection of large vessel occlusion (LVO) stroke with a novel blood test can accelerate the time from triage assessment to thrombectomy puncture. It will unfold in three phases:

Phase 0 - Baseline Data Collection (3 months): Before the random allocation, all clusters undergo data collection on baseline characteristics and outcome measures to confirm/set a pre-intervention comparison ground. Phase 0 patients will receive the current standard of care. An interim analysis will check recruitment rates and explore the need for additional clusters for adequate study power.

Phase 1 - Intervention and Control (12 months): Clusters are randomized to either the intervention or control group, with the intervention arm implementing the LVOne test and the control arm continuing standard care without the LVOne test. Data analysts remain blinded to group allocation, while an interim analysis revisits recruitment and primary outcomes to assess whether additional clusters are required.

Phase 2 - Crossover (12 months): Clusters switch roles from Phase 1, allowing every cluster to experience both the intervention and control conditions, facilitating within-cluster comparisons. The nature of the intervention prevents the blinding of participants and staff.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21 to 85 years old
* Language: Speak and understand Spanish or English
* Residence: Resident of Puerto Rico
* Clinical presentation: Suspected acute stroke
* Time of presentation: Monday to Friday, between 8:00 a.m. and 4:00 p.m.
* Time of symptom onset: symptoms are known to have begun within the last 6 hours, OR last known to be well between 6 and 18 hours ago, confirmed by a reliable witness or healthcare professional

Exclusion Criteria:

* Previous healthcare encounter:
* Already assessed at another hospital, and ambulance admission is a transfer for continuing care OR
* Received thrombolysis therapy before consent (e.g., tPA, alteplase)
* Medical History: diagnosed with any of the following in the past 4 weeks: deep vein thrombosis (DVT), pulmonary embolism (PE), arterial embolism, stroke, transient ischemic attack (TIA), long bone fracture, major trauma, surgery under general anesthesia, or head injury requiring hospital admission within the last 4 weeks.
* Modified Rankin Scale: Pre-stroke mRS ≥ 3
* The patient is a pregnant woman
* The patient is under legal custody or deprived of liberty in penitentiary institutions
* The patient is unable to provide informed consent on their own and whose authorized legal representatives are unavailable in person or by telephone during recruitment

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in the time from triage assessment to thrombectomy puncture | 24 hours
  The difference in time from the participant triage assessment to thrombectomy puncture.

SECONDARY OUTCOMES:
Time from spoke hospital triage assessment to LVOne test in intervention | 24 hours
  Difference in time from triage assessment to the performance of the LVOne test in the intervention group.
Time from HUB hospital triage assessment to LVOne test in intervention | 24 hours
  The difference in time from the HUB hospital triage assessment to the performance of the LVOne test.
Time from HUB hospital triage assessment to thrombectomy puncture | 24 hours
  The difference in time from the HUB hospital triage assessment to the thrombectomy puncture.
Thrombectomy rate (proportion of treated LVO) | 24 hours
  The number of participants that received thrombectomy.
Length of hospital stay | From date of randomization until the date of discharge or date of death from any cause while patient is in hospital, whichever came first, assessed up to 30 days
  The participant's hospitalization period.
Length of ICU stay | From date of randomization until the date of discharge or date of death from any cause while patient is in hospital, whichever came first, assessed up to 30 days
  The participant's hospitalization period in the intensive care unit (ICU).
Diagnostic accuracy for LVO detection | At the time of initial assessment and confirmed by diagnostic imaging within 24 hours
  The ability of the test to correctly identify large vessel occlusion (LVO) in patients with suspected acute ischemic stroke. Diagnostic accuracy will be assessed by comparing the test results to the reference imaging standards.
Diagnostic accuracy for intracerebral hemorrhage detection | At the time of initial assessment and confirmed by diagnostic imaging within 24 hours
  The ability of the LVOne test to correctly detect intracerebral hemorrhage (ICH) in patients presenting with acute stroke symptoms. Diagnostic accuracy will be determined by comparing LVOne test results to diagnostic imaging.
Modified Rankin Scale (mRS) | At the time of initial assessment, 24 hours, at discharge, 3 months, 6 months, and 12 months
  The modified Rankin Scale (mRS) is a measure of functional outcome assessing the degree of disability or dependence in daily activities. The scale ranges from 0 (no symptoms) to 6 (death).

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Vicenty Padilla, MD, Principal Investigator — University of Puerto Rico Medical Sciences Campus
Locations (1):
- Hospital Menonita Caguas, Caguas, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malhotra K, Gornbein J, Saver JL. Ischemic Strokes Due to Large-Vessel Occlusions Contribute Disproportionately to Stroke-Related Dependence and Death: A Review. Front Neurol. 2017 Nov 30;8:651. doi: 10.3389/fneur.2017.00651. eCollection 2017. PMID 29250029
- [Background] Victor P, Bian E, Mamdouh H, Mohamed GA, Nour HA, Miller K, Singh K, Patel S, Segovis C, Nahab F. Upfront vascular imaging in acute stroke: Impact on thrombectomy transfer time at a primary stroke center. J Stroke Cerebrovasc Dis. 2024 Aug;33(8):107815. doi: 10.1016/j.jstrokecerebrovasdis.2024.107815. Epub 2024 Jun 13. PMID 38878844
- [Background] Saver JL. Time is brain--quantified. Stroke. 2006 Jan;37(1):263-6. doi: 10.1161/01.STR.0000196957.55928.ab. Epub 2005 Dec 8. PMID 16339467
- [Background] Durrani Y, Gerstl JVE, Murphy D, et al. Prospective Validation of Glial Fibrillary Acidic Protein, d -Dimer, and Clinical Scales for Acute Large-Vessel Occlusion Ischemic Stroke Detection . Stroke: Vascular and Interventional Neurology. Published online May 17, 2024. doi:10.1161/svin.123.001304
- [Background] Gaude E, Nogueira B, Ladreda Mochales M, Graham S, Smith S, Shaw L, Graziadio S, Ladreda Mochales G, Sloan P, Bernstock JD, Shekhar S, Gropen TI, Price CI. A Novel Combination of Blood Biomarkers and Clinical Stroke Scales Facilitates Detection of Large Vessel Occlusion Ischemic Strokes. Diagnostics (Basel). 2021 Jun 22;11(7):1137. doi: 10.3390/diagnostics11071137. PMID 34206615
- [Background] Kothari RU, Brott T, Broderick JP, Barsan WG, Sauerbeck LR, Zuccarello M, Khoury J. The ABCs of measuring intracerebral hemorrhage volumes. Stroke. 1996 Aug;27(8):1304-5. doi: 10.1161/01.str.27.8.1304. PMID 8711791
- [Background] Puetz V, Dzialowski I, Hill MD, Subramaniam S, Sylaja PN, Krol A, O'Reilly C, Hudon ME, Hu WY, Coutts SB, Barber PA, Watson T, Roy J, Demchuk AM; Calgary CTA Study Group. Intracranial thrombus extent predicts clinical outcome, final infarct size and hemorrhagic transformation in ischemic stroke: the clot burden score. Int J Stroke. 2008 Nov;3(4):230-6. doi: 10.1111/j.1747-4949.2008.00221.x. PMID 18811738
- [Background] Bamford J. Clinical examination in diagnosis and subclassification of stroke. Lancet. 1992 Feb 15;339(8790):400-2. doi: 10.1016/0140-6736(92)90085-h. No abstract available. PMID 1346666
- [Background] van Swieten JC, Koudstaal PJ, Visser MC, Schouten HJ, van Gijn J. Interobserver agreement for the assessment of handicap in stroke patients. Stroke. 1988 May;19(5):604-7. doi: 10.1161/01.str.19.5.604. PMID 3363593
- [Background] Barber PA, Demchuk AM, Zhang J, Buchan AM. Validity and reliability of a quantitative computed tomography score in predicting outcome of hyperacute stroke before thrombolytic therapy. ASPECTS Study Group. Alberta Stroke Programme Early CT Score. Lancet. 2000 May 13;355(9216):1670-4. doi: 10.1016/s0140-6736(00)02237-6. PMID 10905241
- [Background] Goyal M, Fargen KM, Turk AS, Mocco J, Liebeskind DS, Frei D, Demchuk AM. 2C or not 2C: defining an improved revascularization grading scale and the need for standardization of angiography outcomes in stroke trials. J Neurointerv Surg. 2014 Mar;6(2):83-6. doi: 10.1136/neurintsurg-2013-010665. Epub 2013 Feb 6. No abstract available. PMID 23390038
- [Background] Menon BK, Smith EE, Modi J, Patel SK, Bhatia R, Watson TW, Hill MD, Demchuk AM, Goyal M. Regional leptomeningeal score on CT angiography predicts clinical and imaging outcomes in patients with acute anterior circulation occlusions. AJNR Am J Neuroradiol. 2011 Oct;32(9):1640-5. doi: 10.3174/ajnr.A2564. Epub 2011 Jul 28. PMID 21799045